CLINICAL TRIAL: NCT04754529
Title: Influence of Yoga on Cancer-Related Stress in Cancer Survivors
Brief Title: Yoga Intervention for the Improvement of Cancer-Related Stress in Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: I 891720; NCI-2021-00698 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 891720 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2021-02-08; First posted 2021-02-15 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (yoga) (Experimental): Patients receive online yoga intervention QW for 12 weeks.
  Interventions: Other: Quality-of-Life Assessment; Other: Survey Administration; Other: Yoga

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Survey Administration — Ancillary studies
Other: Yoga — Receive yoga intervention
  Other Names: Yoga Therapy

SUMMARY:
This clinical trial develops and test a yoga intervention in improving cancer-related stress in cancer survivors. The online hatha yoga intervention of breathing and movement incorporates both restorative poses, breathing techniques, guided meditation and may reduce stress levels and improve overall quality of health in cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To develop and test the feasibility of a standardized 12-week online hatha yoga intervention (n=30) of breathing and movement incorporating both restorative poses, breathing techniques, guided meditation.

SECONDARY OBJECTIVES:

I. To evaluate the yoga intervention in relation to self-reported levels of stress and quality of life in cancer survivors (n=30).

II. Feasibility of collecting blood and saliva at baseline and post-intervention for stress biomarkers, including cortisol and norepinephrine.

EXPLORATORY OBJECTIVE:

I. To determine how behavior change, quality of life (QoL), and biomarkers of adrenergic stress, inflammation, and immunosuppression are affected by a 12-week online yoga program completed by cancer survivors.

OUTLINE:

Patients receive online yoga intervention once a week (QW) for 12 weeks.

After completion of study, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years of age
* Have been diagnosed with a cancer and have finished treatment
* Have been cleared for physical activity by a physician or nurse practitioner (physician or nurse practitioner name and date clearance received)
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Unwilling or unable to complete the assessment in English
* Are pregnant or nursing
* Are unwilling or unable to follow protocol requirements
* Have skeletal instabilities and/or cardio-pulmonary comorbidities
* Have any condition which in the investigator's opinion deems the subject an unsuitable candidate to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who participate or show high adherence to the intervention | Up to 12 weeks
  Will be presented as observed proportion and 95% Clopper-Pearson confidence intervals (CIs).

SECONDARY OUTCOMES:
Efficacy of the intervention in stress-reduction | Up to 3 months post-intervention
  Serum cortisol and norepinephrine levels will be measured by blood collection
Efficacy of the intervention in stress-reduction | Up to 3 months post intervention
  Self report stress
Efficacy of the intervention in stress reduction | Up to 3 months post intervention
  salivary cortisol will be measured by saliva collection

OTHER OUTCOMES:
Change in Quality of life | Up to 3 months post-intervention
  Quality of life collected by the EORTC Quality of Life Questionnaire
Change in Cognitive function | Up to 12 weeks
  Cognitive function will be assessed by standard questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Glaser, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States